CLINICAL TRIAL: NCT05639270
Title: Pilot Study Before/After of Vagal Stimulation in Chronic Low Back Pain
Brief Title: Pilot Study of Vagal Stimulation in Chronic Low Back Pain
Acronym: VALOM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL21_0598
Record Dates: First submitted 2022-11-28; First posted 2022-12-06 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-02

CONDITIONS: Low Back Pain
Keywords: Vagus nerve stimulation; low back pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- low back pain (Experimental): The experimental intervention consists of vagal stimulation using the Tens Eco device with an auricular electrode and conductive gel.
  The stimulation will have an intensity of 25 Hz, lasting 30 minutes, once a day, for 3 months.
  An evaluation of the pain will be done every week by phone for the first month and then in consultation at one month and at 3 months.
  Interventions: Device: use of an auricular electrode

INTERVENTIONS:
Device: use of an auricular electrode — Use of the auricular electrode throughout the duration of the study (30minutes/day) combined with assessment of pain, tolerance, vagal tone.

SUMMARY:
Low back pain is a major public health problem. It is the leading cause of disability in the world. The factors that lead to chronicity of low back pain are multi-factorial and are essentially represented by psychosocial factors (catastrophism, kinesiophobia, algophobia job dissatisfaction, emotional problems such as depression, anxiety, stress, injustice, etc.).

Pain is a multimodal experience that involves different brain structures that are activated by the pain signal and involve the autonomic nervous system (ANS). The vagus nerve is the main actor of one of the two branches of the ANS, the parasympathetic system, which acts as a "slow-down".

The vagus nerve participates in the inter-neuronal transmission of key neurotransmitters for mood, alertness, attention and motivation.

Vagal stimulation has been used for many years as an analgesic device in chronic pain (vascular pain (facial vascular pain, fibromyalgia, visceral pain, gastrointestinal and pelvic pain...)

To date, no study has been conducted on the value of vagal stimulation in chronic low back pain.

DETAILED DESCRIPTION:
Low back pain is a major public health problem. It is the leading cause of disability in the world.

The factors that lead to chronicity of low back pain are multifactorial, which explains the modest effectiveness of both drug treatments and multidisciplinary programs (analgesic drug interventions, non-pharmacological interventions with rehabilitation, physical exercise, psychotherapy, spinal ergonomics, meditation, yoga, etc.) in the treatment of low back pain. psychotherapy, spinal ergonomics, meditation, yoga...) in chronic forms. These factors of chronicization are essentially represented by psychosocial factors (catastrophism, kinesiophobia, algophobia, job dissatisfaction, emotional problems such as depression, anxiety stress, injustice...)

In the chronic low back pain population, pain is a multimodal experience that involves different brain structures (insula, anterior cingulate cortex, amygdala and prefrontal cortex). These structures are activated by the pain signal and involve the autonomic nervous system (ANS).

The vagus nerve is the main actor of one of the two branches of the ANS, the parasympathetic system, which acts as a "slow-down".

The vagus nerve is involved in the inter-neuronal transmission of key neurotransmitters for mood, alertness, attention and motivation (serotonin, dopamine, oxytocin and noradrenaline).

It is one of the longest nerves in the human body, originating from the base of the brain (nucleus tractus solitarius) and innervating most of the organs (heart, lung, stomach, liver, spleen, kidneys, gallbladder, pancreas, intestines). It allows the integration of information from the periphery (pain, stress, emotions), slows down the heart rate after a stress, reduces the caliber of the bronchial tubes to help breathing, reduces the inflammatory response, participates in digestion and in the communication with the digestive microbiota.

Indeed, there seems to be an alteration of the vagal function in chronic pain patients patients: the vagus nerve is involved in the modulation of pain at different levels (medullary, cerebral) (medullary, cerebral) but also on the different components of pain (sensory, affective emotional, behavioral).

The benefit of the stimulation of the vagus would be mediated by a modulation of afferent information (stress, pain, emotion) associated with a benefit of "relaxation" conveyed by the efferent fibers (cardiac, pulmonary effect...).

This stimulation of the vagus nerve is done through an atrial electrode that stimulates the atrial branch of the vagus nerve.

To date, no study has been conducted on the value of vagal stimulation in chronic low back pain.

Because of the multifactorial mechanisms involved in this pathology, this type of therapy appears to be a useful complement to the management of our patients.

This pilot study will allow us to evaluate the feasibility of a larger study with a placebo arm.

The evaluation of tolerance and adherence to this therapy will be taken into account.

ELIGIBILITY:
Inclusion Criteria:

* Low back pain with a VAS greater than or equal to 40 that has been ongoing for more than 3 months
* Failed or insufficiently relieved by private physiotherapy
* Failed or insufficiently relieved or intolerant of level II analgesics
* No change in therapy envisaged within one month.

Exclusion Criteria:

* Non-common low back pain will not be accepted (presence of red flags).
* Auricular canal not adapted to the stimulation device.
* Use of another type of electrical device (pacemaker or TENS).
* History of vagotomy.
* Heart rhythm disorder.
* Presence of a cochlear implant on the stimulation side
* Pregnancy in progress or planned during the study period
* Adult protected by law or patient under guardianship or curator
* Person unable to give consent.
* Participation in other ongoing biomedical research
* Absence of express informed consent after a reflection period
* Not being affiliated to a French social security system or being a beneficiary of such a system

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
change from baseline pain at 1 month | between baseline and 1 month
  evaluated by a Visual Analog Scale (VAS, 0 the worst result and 100 the best result)

SECONDARY OUTCOMES:
change from baseline functional disability at 1 month | between baseline and 1 month
  evaluated by Oswestry score The questionnaire consists of 10 questions, concerning: pain, self-care, load carrying, walking, sitting, standing, sleep, sexual life, social life, travel.
  Score between 0 and 20%: minimal disability Score between 21 and 40%: moderate disability Score between 41 and 60% : severe disability Score between 61 and 80% : major disability Score between 81 and 100% : bedridden patient
change from baseline functional disability at 3 month | between baseline and 3 month
  evaluated by Oswestry score The questionnaire consists of 10 questions, concerning: pain, self-care, load carrying, walking, sitting, standing, sleep, sexual life, social life, travel.
  Score between 0 and 20%: minimal disability Score between 21 and 40%: moderate disability Score between 41 and 60% : severe disability Score between 61 and 80% : major disability Score between 81 and 100% : bedridden patient
change from baseline quality of life at 1 month | between baseline and 1 month
  evaluated by EQ-5D-5L score (0 to 20, 0 the better, and 20 the worst ; 0 to 100 for the L part, 0 the worst and 100 the better)
change from baseline quality of life at 3 month | between baseline and 3 month
  evaluated by EQ-5D-5L score (0 to 20, 0 the better, and 20 the worst ; 0 to 100 for the L part, 0 the worst and 100 the better)
change from baseline anxiety and depression at 1 month | between baseline and 1 month
  evaluated by HAD (Hospital Anxiety and Depression scale) score
change from baseline anxiety and depression at 3 month | between baseline and 3 month
  evaluated by HAD (Hospital Anxiety and Depression scale) score
change from baseline catastrophism at 1 month | between baseline and 1 month
  evaluated by PCS (Pain Catastrophizing Scale) score
change from baseline catastrophism at 3 month | between baseline and 3 month
  evaluated by PCS (Pain Catastrophizing Scale) score
evolution of use of painkillers at 1 month | between baseline and 1 month
evolution of use of painkillers at 3 month | between baseline and 3 month
evaluation of device adherence at 1 month | between baseline and 1 month
  number of stimulations performed
evaluation of device adherence at 3 month | between baseline and 3 month
  number of stimulations performed
evaluation of device tolerance at 1 month | between baseline and 1 month
  number of adverse events
evaluation of device tolerance at 3 month | between baseline and 3 month
  number of adverse events
evaluation of device satisfaction at 1 month | between baseline and 1 month
  Lickert scale from 1 to 5.
evaluation of device satisfaction at 3 month | between baseline and 3 month
  Lickert scale from 1 to 5.
change from baseline vagal tone at 1 month | between baseline and 1 month
  evaluated by Heart Rate variability
change from baseline vagal tone at 3 month | between baseline and 3 month
  evaluated by Heart Rate variability

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU Montpellier, Montpellier
  - CHU Nîmes - Le Grau du Roi, Nîmes